CLINICAL TRIAL: NCT04615689
Title: The Association of Gut Microbiota With Urinary Tract Infection in Infants
Status: Withdrawn | Type: Observational
Why Stopped: Because of the covid 19 pandemic, no patients were enrolled.
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Ky Young Cho, Associate Professor, Hallym University Kangnam Sacred Heart Hospital
Other Study IDs: Gut microbiota and UTI
Record Dates: First submitted 2020-10-23; First posted 2020-11-04 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigators will sequence the V3-V4 of the bacterial 16SrRNA genes from the feces.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infants with febrile urinary tract infection: The investigators will recruit infants hospitalized for acute febrile urinary tract infection. Before starting antibiotics treatment, The investigators will collect feces with the informed consents from infants' parents.
  Interventions: Other: The collection of feces
- Healthy infants: The investigators will recruit healthy controls from the clinics for routine check up with the informed consents from infants' parents.
  Interventions: Other: The collection of feces

INTERVENTIONS:
Other: The collection of feces — When the infants will be diagnosed with urinary tract infection, feces will be collected. Feces will be collected from healthy infants with informed consent.

SUMMARY:
This prospective case-control study will compare the gut microbiota between the infants with febrile urinary tract infection and healthy infants.

DETAILED DESCRIPTION:
The investigators hypothesize that the gut environment reflected by intestinal microbiota influences the risk of urinary tract infection. This prospective case-control study will compare the gut microbiota between the infants with febrile urinary tract infection and healthy infants. The investigators will sequence the V3-V4 of the bacterial 16SrRNA genes from the feces and analyze the sequencing data by QIIME2.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of febrile urinary tract infection.
* Infants

Exclusion Criteria:

* Congenital kidney disease
* Congenital heart disease
* Other metabolic disease

Ages: 6 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants hospitalized for febrile urinary tract infection. Healthy controls who visited at primary care clinic for routine check up with informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
The differential compositional analysis of the gut microbiota between healthy controls and infants with febrile urinary tract infection. | An average of 1 year, after the completion of recruitment.
  The investigators will sequence the V3-V4 of the bacterial 16SrRNA genes from the feces and analyze the sequencing data by QIIME2. From the OTU table, the investigators will conduct the differential compositional analysis of the gut microbiota between healthy controls and infants with febrile urinary tract infection, using the linear discriminant analysis and analysis of differential abundance taking sample variation into account in R program and QIIME2.

SECONDARY OUTCOMES:
The differential functional analysis of the gut microbiota between healthy controls and infants with febrile urinary tract infection. | An average of 1 year, after the completion of recruitment.
  The investigators will predict the functional analysis from the OTU table and compare those results between healthy controls and infants with febrile urinary tract infection, using PICRUST2 analysis.

CONTACTS AND LOCATIONS:
Overall Officials: KY YOUNG CHO, M.D, Ph.D, Principal Investigator — Hallym University Kangnam Sacred Heart Hospital
Locations (1):
- Hallym University Kangnam Sacred Heart Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No